CLINICAL TRIAL: NCT04540874
Title: Safety, Tolerability and Pharmacokinetics of Single Rising Oral Doses of BI 894416 Versus Placebo in Healthy Male Japanese Subjects (Single-blind, Randomized, Placebo-controlled Within Dose Group)
Brief Title: A Study in Healthy Japanese Men to Test How Different Doses of BI 894416 Are Tolerated
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: due to company decision
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1371-0003
Record Dates: First submitted 2020-09-04; First posted 2020-09-07 (Actual); Results first posted 2023-08-16 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2022-09

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BI 894416 25mg (Experimental): 1 tablet of 25 milligrams (mg) BI 894416 was administered orally as single dose with 240 milliliters of water after an overnight fast of at least 10 hours on day 1, followed by at least 48 hours close medical surveillance, followed by 2 weeks of follow-up period.
  Interventions: Drug: BI 894416
- Placebo group (Placebo Comparator): Matching placebo was administered orally as single dose with 240 milliliters of water after an overnight fast of at least 10 hours on day 1, followed by at least 48 hours close medical surveillance, followed by 2 weeks of follow-up period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BI 894416 — BI 894416
  Arms: BI 894416 25mg
Drug: Placebo — Placebo
  Arms: Placebo group

SUMMARY:
The objective of this trial is to investigate the safety, tolerability and pharmacokinetics of BI 894416 in healthy Japanese male subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male subjects according to the assessment of the investigator, as based on a complete medical history, including a medical examination, vital signs (Blood pressure (BP), Pulse rate (PR)), 12-lead Electrocardiogram (ECG), and clinical laboratory tests
2. Japanese ethnicity, according to the following criteria:

   - born in Japan, have lived outside of Japan <10 years, and have parents and grandparents who are Japanese
3. Age of 20 to 45 years (inclusive) at screening
4. BMI of 18.5 to 25.0 kg/m2 (inclusive) at screening
5. Signed and dated written informed consent prior to admission to the trial, in accordance with Good Clinical Practice (GCP) and local legislation
6. Subjects who agree to minimize the risk of making their partner pregnant by fulfilling any of the following criteria starting from the first administration of trial medication until 90 days after last administration of trial medication

   * Use of adequate contraception, any of the following methods plus condom:

intrauterine device, combined oral contraceptives that started at least 2 months prior to the first drug administration

* Vasectomized (vasectomy at least 1 year prior to enrolment)
* Surgical sterilization (including bilateral tubal occlusion, hysterectomy or bilateral oophorectomy) of the subject's female partner

Exclusion Criteria:

1. Any finding in the medical examination (including BP, PR or ECG) deviating from normal and assessed as clinically relevant by the investigator
2. Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 50 to 90 bpm
3. Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
4. Any evidence of a concomitant disease assessed as clinically relevant by the investigator
5. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
6. Cholecystectomy or other surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication, except appendectomy or simple hernia repair
7. Diseases of the central nervous system, including but not limited to, any kind of seizures or stroke, and other relevant neurological or psychiatric disorders
8. History of relevant orthostatic hypotension, fainting spells, or blackouts Further exclusion criteria apply.

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2020-10-05 (Actual); Primary Completion 2020-11-12 (Actual); Study Completion 2020-11-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Research Hospital Tokyo, Tokyo, Shinjuku-ku, Japan

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions:
  1. studies in products where Boehringer Ingelheim is not the license holder; 2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; 3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization).
  For more details refer to: http://trials.boehringer-ingelheim.com/

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This single-blind, randomised, placebo-controlled within dose group study investigated the safety, tolerability, and pharmacokinetics of single rising oral doses of BI 894416 versus placebo in healthy male Japanese subjects followed by 48 hours close medical surveillance and 2 weeks of follow-up period thereafter. This trial was prematurely terminated due to decision of sponsor.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria.
  Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Groups:
- Placebo: Matching placebo was administered orally as single dose with 240 milliliters of water after an overnight fast of at least 10 hours on day 1, followed by at least 48 hours close medical surveillance, followed by 2 weeks of follow-up period.
Period: Overall Study
Arm/Group | BI 894416 25mg | Placebo
Started | 6 | 2
Completed | 6 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS): The treated set includes all subjects who were randomized and treated with at least one dose of investigational medicinal product. The treatment assignment will be determined based on the first treatment the subjects received.
Groups:
- Total: Total of all reporting groups
Arm/Group | BI 894416 25mg | Placebo | Total
Number analyzed (Participants) | 6 | 2 | 8
Age, Continuous [Mean (Standard Deviation); unit: Years] | 31.5 (7.7) | 31.5 (12.0) | 31.5 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 6 | 2 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 2 | 8
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 6 | 2 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Drug Related Adverse Events
Description: The percentage of participants with drug related adverse events was reported.
Time Frame: From drug administration until end of follow-up, up to 17 days.
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants
Arm/Group | BI 894416 25mg | Placebo
Number analyzed (Participants) | 6 | 2
Percentage of participants | 16.7 | 0.0

2. Secondary Outcome: Area Under the Concentration-time Curve of BI 894416 in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-∞)
Description: Area under the concentration-time curve of BI 894416 in plasma over the time interval from 0 extrapolated to infinity was reported.
Time Frame: Within 1 hour (h) before drug administration and at 15 minutes (min), 30min, 45min, 1h, 1h30min, 2h, 2h30min, 3h, 4h, 5h, 6h, 8h, 10h, 12h, 24h, 34h, 48h, 72h after drug administration.
Population: Pharmacokinetic (PK) parameter analysis set (PKS): This set includes all subjects in the treated set who provide at least one PK endpoint that was not excluded due to a protocol violation relevant to the evaluation of PK or due to PK non-evaluability. Thus, a subject will be included in the PKS, even if he contributes only one PK parameter value for one period to the statistical assessment.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour * nanomole / liter
Arm/Group | BI 894416 25mg
Number analyzed (Participants) | 6
hour * nanomole / liter | 3550 (26.6)

3. Secondary Outcome: Maximum Measured Concentration of BI 894416 in Plasma (Cmax)
Description: Maximum measured concentration of BI 894416 in plasma was reported.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomole / liter
Arm/Group | BI 894416 25mg
Number analyzed (Participants) | 6
nanomole / liter | 708 (25.0)

ADVERSE EVENTS:
Time Frame: From drug administration until end of follow-up, up to 17 days.
Description: Treated set (TS): The treated set includes all subjects who were randomized and treated with at least one dose of investigational medicinal product. The treatment assignment will be determined based on the first treatment the subjects received.
Groups:
- Total: All treated participants in this study.
Arm/Group | BI 894416 25mg | Placebo | Total
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/2 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/2 | 0/8
Other Adverse Events (participants affected / at risk) | 1/6 | 1/2 | 2/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BI 894416 25mg (N=6) | Placebo (N=2) | Total (N=8)
Feeling abnormal (General disorders) | 1 | 0 | 1
Blood triglycerides increased (Investigations) | 0 | 1 | 1

LIMITATIONS AND CAVEATS:
The study was terminated by the sponsor after the first dosage group (25 mg BI 894416), only a subset of the analyses planned in the protocol was performed. No dose-proportionality analysis was done. Secondary endpoints were analysed descriptively only.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results.

Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days.

BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2020-08-17): https://cdn.clinicaltrials.gov/large-docs/74/NCT04540874/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-12): https://cdn.clinicaltrials.gov/large-docs/74/NCT04540874/SAP_001.pdf